CLINICAL TRIAL: NCT06627517
Title: Automated Insulin Delivery for Multiple Daily Injectors (AID4MDI)
Brief Title: Safety and Effectiveness of the Luna System in People With Type 1 Diabetes Mellitus
Acronym: AID4MDI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Luna Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LH2024-01
Record Dates: First submitted 2024-10-02; First posted 2024-10-04 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2024-12

CONDITIONS: Type 1 Diabetes Mellitus; Sleep Quality
Keywords: overnight hyperglycemia; sleep quality; type 1 diabetes; closed loop
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Overnight wear of study device (Experimental): Subjects will wear the study device during sleep in addition to their usual basal/bolus therapy.
  Interventions: Device: Episodic overnight patch pump

INTERVENTIONS:
Device: Episodic overnight patch pump — Subjects will wear the study device overnight for a period of 13 weeks in conjunction with use of Dexcom G6.

SUMMARY:
The purpose of this research is to evaluate the effect of a wearable insulin pump on blood sugar levels during sleep. The study device works with continuous glucose monitors (CGM) to calculate and deliver rapid-acting insulin doses during sleep. The study device does not replace long-acting, correction, or mealtime insulin. The study will involve applying the study device before bed for a period of 13 weeks. The overall study length is approximately 17 weeks.

The study aims to evaluate whether the study device is safe and if it lowers blood sugar levels in people who have consistently high blood sugar during sleep and at wake.

ELIGIBILITY:
Inclusion Criteria

1. ≥18 years of age at time of consent
2. Clinical diagnosis of T1D for ≥ 6 months with a stable insulin regimen for ≥ 30 days.
3. Using a basal-bolus regimen with multiple daily injections of insulin or doses of inhaled insulin for ≥ 3 months with a stable basal dosing regimen over the previous 30 days
4. If using a non-insulin glucose-lowering drug, (e.g. GLP-1 agonists, SGLT2 inhibitors), must have a stable dose for ≥ 30 days
5. If using a weight loss medication, must be on a stable dose for ≥ 30 days
6. Using insulin lispro or insulin aspart as bolus insulin or able to obtain for the duration of the study

5. If using a weight loss medication, must be on a stable dose for ≥ 30 days 6. Using insulin lispro or insulin aspart as bolus insulin or able to obtain for the duration of the study 7. Using CGM (real-time or intermittent scanning) for ≥ 3 months (with at least 50% use), and at least 85% use in the prior 14 days 8. Using Dexcom G6 or able to obtain for the duration of the study 9. Using an iPhone as part of daily life or able to obtain for the duration of the study 10. Recurrent nocturnal hyperglycemia, defined as ≥ 7 of the previous 14 days with a nighttime glucose value > 180 mg/dL.

* Nighttime is defined at the discretion of the investigator and is intended to be the time period from when the subject goes to bed to when they get up in the morning 11. Negative baseline pregnancy test. Females of childbearing potential, willing to use an adequate method of birth control for the duration of the study.
* Adequate methods of birth control include hormonal contraceptives, intrauterine devices, or double barrier contraception, e.g., condom + diaphragm, condom or diaphragm + spermicidal gel, or foam.
* Menopause is defined as one year without menses; if in question, a follicle stimulating hormone of >40 U/ml must be documented.
* Hysterectomy, bilateral oophorectomy, or bilateral tubal ligation must be documented as applicable.

  12. Availability of a relative or acquaintance residing within 15 minutes of the subject and willing to be the subject's care partner throughout the study.
* The care partner must be willing to be trained on how to use the Dexcom Follow app and administer glucagon.
* The care partner must be willing to contact the subject upon a low or high alarm, provide aid to the subject, including glucagon administration, and/or contact emergency services.

  13. Willing to share access to CGM data with the Sponsor through the Dexcom Clarity app 14. No medical, psychiatric, or other conditions, or medications being taken that in the Investigator's judgement would be a safety concern for participation in the study. This includes considering the potential impact of medical conditions known to be present including cardiovascular, liver, kidney disease, thyroid disease, adrenal disease, malignancies, vision difficulties, active proliferative retinopathy, and other medical conditions; psychiatric conditions including eating disorders; drug or alcohol abuse.

Exclusion Criteria

1. Use of or plan to use insulin pump therapy during the study period.
2. Use of basal insulin for ≥ 60% of the total daily insulin dose on average over the last week per subject report.
3. Pregnant, lactating, or plans to become pregnant in the next 17 weeks. A negative serum or urine pregnancy test is required for all females of child-bearing potential.
4. Known stage 4/5 renal failure or on dialysis
5. Using Hydroxyurea medication
6. Current or anticipated acute use of corticosteroids (other than topical or inhaled) or other medications that have a known effect on glycemic variability during the time period of the study
7. Anticipated initiation of a weight loss medication and/or titration during the study period
8. Alcohol or drug use that would reduce sensitivity to symptoms of hypoglycemia or hinder appropriate decision-making in the judgment of the investigator.
9. Use of electrically powered implant(s) that may be susceptible to RF interference, such as cardiac pacemakers, spinal cord stimulators, or implantable cardioverter-defibrillators.
10. Severe hypoglycemia (defined as requiring 3rd party assistance and/or loss of consciousness or seizure) within 90 days prior to screening.
11. Diabetic ketoacidosis (DKA) diagnosed at a health care facility within 90 days prior to screening
12. Use of an investigational drug in the 30 days prior to screening.
13. Employed by or has immediate family members employed by Luna Health; is directly involved in conducting the clinical study; has a direct supervisor at the place of employment who is also directly involved in conducting the clinical study (as a study investigator, coordinator, etc.); or has a first-degree relative who is directly involved in conducting the clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Severe hypoglycemia events | From device activation to the end of treatment at 13 weeks
Diabetic ketoacidosis events | From device activation to the end of treatment at 13 weeks
Change in CGM-measured time in range (70-180 mg/dL) | From device activation to the end of treatment at 13 weeks

SECONDARY OUTCOMES:
Change in CGM-measured percentage of time > 180 mg/dL | From device activation to the end of treatment at 13 weeks
Change in CGM-measured percentage of time > 250 mg/dL | From device activation to the end of treatment at 13 weeks
Change in CGM-measured percentage of time waking in range (70-180 mg/dL) | From device activation to the end of treatment at 13 weeks
Change in CGM-measured fasting glucose at the end of the sleep period | From device activation to the end of treatment at 13 weeks
Change in Pittsburgh Sleep Quality Index (PSQI) score | From device activation to the end of treatment at 13 weeks
  Scale of 0 to 21 with higher scores being a worse outcome
Change in HbA1c | From device activation to the end of treatment at 13 weeks
Change in Epworth Sleepiness Scale (ESS) score | From device activation to the end of treatment at 13 weeks
  Scale of 0 to 24 with higher scores being a worse outcome
Rate, severity, and device-relatedness of all adverse events | From device activation to the end of treatment at 13 weeks
Change in CGM-measured time < 70 mg/dL | From device activation to the end of treatment at 13 weeks
Change in CGM-measured time < 54 mg/dL | From device activation to the end of treatment at 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy H Pettus, MD, Principal Investigator — University of California, San Diego
Locations (3):
- United States (3):
  - Diablo Clinical Research, Walnut Creek, California
  - Barbara Davis Center for Diabetes, Aurora, Colorado
  - International Diabetes Center, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: Yes